CLINICAL TRIAL: NCT05903638
Title: A Pilot RCT: the Impact of a Virtual MBSR Course on Women With Primary Infertility Seeking Fertility Treatment at a Single Centre
Brief Title: A Pilot RCT: the Impact of a Virtual MBSR Course on Women With Primary Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: One Fertility (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MBSR Pilot RCT
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Primary Infertility; Mental Health Issue; Quality of Life

STUDY DESIGN:
Intervention Model Description: Single-blinded pilot randomized control trial with control arm and intervention (virtual MBSR course).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Virtual Mindfulness-Based Stress Reduction (MBSR) program (Experimental)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction course

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction course — 8-week, 26-hour, virtual mindfulness course
  Other Names: MBSR
  Arms: Virtual Mindfulness-Based Stress Reduction (MBSR) program

SUMMARY:
We plan to perform a pilot study in which women with primary infertility seeking an initial fertility consultation will be randomized into either a standard treatment group or an 8-week virtual Mindfulness-Based Stress Reduction (MBSR) program. Primary outcomes included retention and survey completion rates. Secondary outcomes included Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Perceived Stress Score (PSS), Fertility Problem Index (FPI), pregnancy rates, intention to pursue treatment and % pursuing treatment.

ELIGIBILITY:
Inclusion Criteria:

-Primary infertility and no prior fertility treatment

Exclusion Criteria:

* No internet access
* Non-English speaking
* History of suicidal ideation/intent, psychotic disorder, eating disorder, substance abuse or dependence, PTSD
* Psychotropic medication change in the previous month
* Previously seen at another fertility clinic
* Previous MBSR course
* Previous mindfulness meditation retreat

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
MBSR course participation rate | 8-weeks of MBSR course
Survey completion rate | Randomization to 3-months after course completion

SECONDARY OUTCOMES:
Beck Depression Inventory | Randomization to 3-months after course completion
Beck Anxiety Inventory | Randomization to 3-months after course completion
Perceived Stress Scale | Randomization to 3-months after course completion
Fertility Problem Inventory | Randomization to 3-months after course completion
% involvement in fertility treatment | 3-months after course completion
Pregnancy rates | 3-months after course completion

CONTACTS AND LOCATIONS:
Overall Officials: Mehrnoosh Faghih, MD, Principal Investigator — McMaster University, ONE Fertility
Locations (1):
- ONE Fertility, Hamilton, Ontario, Canada